CLINICAL TRIAL: NCT06383520
Title: Study on the Clinical Application Value of PET Imaging Targeting GPC3 in Hepatocellular Carcinoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0415
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-12

CONDITIONS: Malignant Neoplasm of Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET imaging targeting GPC3 in hepatocellular carcinoma (Experimental): Determine if targeting GPC3 PET is safe and effective method for imaging of hepatocellular carcinoma
  Interventions: Drug: 68Ga-aGPC3-scFv/Fab

INTERVENTIONS:
Drug: 68Ga-aGPC3-scFv/Fab — For pharmacokinetics, healthy volunteer underwent PET imaging targeting GPC3. Blood samples were collected at 25 min, 55 min, and 115 min after imaging agent injection, and urine specimens were collected at 28 min, 58 min, and 118 min after injection to measure radioactivity in blood and urine. PET/MR scans were performed at 30-50 min, 60-80 min, and 120-140 min after injection to understand absorption, distribution, and metabolism.
  For Cancer patients, subjects should have targeting GPC3 and 18F-FDG PET scans two days apart.
  Blood tests, liver and kidney function, tumor markers (AFP, etc.), and other biochemical markers must be performed one week prior to and after imaging.
  Tumor biopsies or surgical specimens should be evaluated histopathologically and immunostained for biomarkers associated with angiogenesis.
  Other Names: gallium-68(68Ga)-aGPC3-scFv/Fab

SUMMARY:
This is a diagnostic study. Patients were recruited from patients with clinically suspected or confirmed hepatocellular carcinoma and healthy volunteers were recruited for PET/or PET/CT imaging targeting a GPC3-specific probe (in the case of 68Ga-NOTA-aGPC3-scFv) , to observe the reaction of volunteers and patients after injection of drugs, to evaluate the pharmacokinetics in vivo and the efficacy of diagnosis and staging, and to perform PET CT imaging in patients with contraindications. General Information, clinical data, blood routine, liver and renal function, and other imaging data were collected. The final diagnosis was based on the histopathology of biopsy or surgical specimens.

DETAILED DESCRIPTION:
Liver cancer is one of the most common malignant tumors in the world, and hepatocellular carcinoma (HCC) is the most prominent histopathological type. Surgical resection and liver transplantation are the main radical methods for early HCC patients. However, due to its insidious onset, more than 90% of HCC patients are already in local advanced stage or accompanied by distant metastasis when diagnosed, so there is no surgical opportunity and the prognosis is very poor. It is important to explore new methods and strategies for early and accurate diagnosis of HCC to improve the prognosis of patients.

Traditional imaging methods such as multi-temporal computed tomography (CT) and magnetic resonance imaging (MRI) have been widely used in the diagnosis, staging and treatment decision making of HCC, but qualitative diagnosis cannot be achieved. Nuclear medicine diagnostic tool [18F]-Fluorodeoxyglucose positron emission tomography/computed tomography ([18F]-FDG PET/CT) imaging technology has been widely used in the diagnosis of a variety of malignant tumors, but due to its low diagnostic accuracy for HCC, especially highly differentiated HCC, its value in the early diagnosis of HCC is limited.

GPC3, a member of the heparan sulfate glycoprotein family, is composed of a core protein, two heparan sulfate chains located at the C-terminal and phosphatidyl inositol anchors attached to the cell membrane. Data analysis showed that GPC3 was significantly overexpressed in tumor cells of HCC patients, but hardly expressed in normal liver tissue or in benign liver diseases, making it the most specific tumor marker for HCC. High expression of GPC3 is associated with poor prognosis in HCC. patients,.suggesting that GPC3 may be an important molecular target for accurate diagnosis and treatment of HCC.

This project proposes to PET imaging targeting GPC3 in the diagnosis and staging of HCC and to compare the diagnostic efficacy with the pathology gold standard. And this study was conducted to compensate for the lack of value of 18F-FDG PET imaging for the diagnosis and staging of malignant tumors by comparing PET imaging targeting GPC3 with the commonly used 18F-FDG PET imaging.

ELIGIBILITY:
Inclusion Criteria:

* 1: Voluntarily participate and the person or their legal representative can sign an informed consent form
* 2: Adult patients (18 years of age or older), regardless of gender
* 3: Patients with newly diagnosed hepatocellular carcinoma with high clinical suspicion or confirmation (supporting evidence including imaging data and histopathologic examination, etc.) who agree to undergo histopathologic examination (if not performed prior to imaging) or/and 18F-FDG PET imaging
* 4: Healthy volunteer
* 5: Patients with a history of hepatocellular carcinoma, remission and recurrence after treatment
* 6: Willing and able to follow schedule visits, treatment plans and laboratory tests

Exclusion Criteria:

* 1: Pregnant or lactating patients
* 2: The patient or their legal representative is unable or unwilling to sign the informed consent form
* 3: Acute systemic diseases and electrolyte disorders
* 4: Patients who are known to be allergic to GPC3 imaging agents or synthetic excipients
* 5: Fasting blood glucose levels exceeding 11.0 mmol/L before injection of 18F-FDG
* 6: Individuals who are unable to complete PET/MR or PET/CT examinations (including inability to lie flat, claustrophobia, radiation phobia, etc.)
* 7: Researchers believe that compliance is poor or there are other unfavorable factors for participating in this experiment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Visual and standardized uptake values assessment of lesions and biodistribution | 1 year
  At least two experienced nuclear medicine physicians will conduct a visual analysis using consensus reading. The standardized uptake value (SUV) of tumor and organs will be measured after a semiquantitative analysis is conducted for each case. The SUV ranges from 0 to infinity, and a higher score means a higher uptake of targeting GPC3 nuclear probe by the tumor, which implies a greater threat of the tumor being malignant or higher stage.

SECONDARY OUTCOMES:
Radioactivity in the blood and urine samples | 1 year
  Blood samples were collected at 25 minutes, 55 minutes and 115 minutes after
Concentration of tumor markers (e.g., APF) in participants' blood | 1 year
  Concentrations of blood tumor markers (e.g., AFP) measured on the date closest to the participant's examination will be collected. A higher blood tumor marker concentration means a higher threat or stage of tumor malignancy.
Pathological sections of tumour tissue | 1 year
  The excised tumour tissue was taken for immunohistochemistry to verify its GPC3 expression

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China